CLINICAL TRIAL: NCT04916197
Title: Effect of Postoperative Prolonged Sedation With Dexmedetomidine After Successful Reperfusion With Endovascular Thrombectomy on Long-term Prognosis in Patients With Acute Ischemic Stroke (PPDET)
Brief Title: Effect of Postoperative Prolonged Sedation With Dexmedetomidine After Successful Reperfusion With EVT on Long-term Prognosis in Patients With AIS (PPDET)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Changwei Wei, Deputy chief physician, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00375929
Record Dates: First submitted 2021-05-25; First posted 2021-06-07 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Acute Ischemic Stroke
Keywords: Endovascular thrombectomy; Dexmedetomidine; Modified Rankin Scale
MeSH Terms: conditions — Ischemic Stroke | interventions — Saline Solution

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Dexmedetomidine 0.1~1.0 μg/kg/h for 24h after patients finished endovascular thrombectomy and returned to ICU. Maintain Ramsay score 2-3.
  Interventions: Drug: Dexmedetomidine prolonged sedation
- Control group (Placebo Comparator): An equal dose of saline 24h after patients finished endovascular thrombectomy and returned to ICU. If the Ramsay sedation score is 1, propofol will be administrated to maintain the Ramsay sedation score at 2 to 3.
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: Dexmedetomidine prolonged sedation — Dexmedetomidine for 24h after patients finished endovascular thrombectomy and returned to ICU.
  Arms: Intervention group
Drug: 0.9% saline — An equal dose of 0.9% saline 24h after patients finished endovascular thrombectomy and returned to ICU.
  Arms: Control group

SUMMARY:
Dexmedetomidine can attenuate the activity of the sympathetic nervous system under stress response and improve ischemia-reperfusion injury. The investigators hypothesized that the prolonged sedation of dexmedetomidine after successful reperfusion of endovascular thrombectomy may improve the clinical outcome of acute ischemic stroke patients.

DETAILED DESCRIPTION:
Endovascular treatment with mechanical thrombectomy is the standard treatment for acute large vessel occlusion.

Dexmedetomidine is a commonly used sedative in endovascular thrombectomy of acute ischemic stroke.

Dexmedetomidine can attenuate the activity of the sympathetic nervous system under stress response and improve ischemia-reperfusion injury.

The investigators hypothesized that the prolonged sedation of dexmedetomidine after successful reperfusion of endovascular thrombectomy may improve the clinical outcome of acute ischemic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* 2≤NIHSS≤25
* mRS score before stroke was less than 3
* Acute ischemic stroke (including anterior circulation)
* mTICI rate 2b or 3
* According to the 2018 AHA/ASA guidelines for the management of acute ischemic stroke, patients who plan to receive mechanical thrombectomy under local anesthesia and sedation
* Informed consent was signed by patient or legal representative

Exclusion Criteria:

* Intracerebral hemorrhage occurred in the responsible vessel area in the past 6 weeks
* Patients who had received stent treatment at the responsible vessel in the past
* Neurological function was restored at or before angiography
* Patients who are allergic to heparin, aspirin, clopidogrel, rapamycin, lactic acid polymer, poly (n-butyl methacrylate), stainless steel, anesthetics and contrast agents or have contraindications
* Hemoglobin was less than 70g/L, platelet count was less than 50×109/L, international normalized ratio (INR) greater than 1.5 (irreversible), there are uncorrectable bleeding factors
* Blood glucose < 2.7 mmol/L or > 22.2 mmol/L
* Severe liver or kidney disfunction, ALT>3 times the upper limit of normal value or AST>3 times the upper limit of normal value, creatinine>1.5 times the upper limit of normal value
* Pregnant or lactating women
* Previous history of mental illness
* Stroke with other acute diseases or postoperative stroke of other operation
* Heart rate less than 50bpm, second or third degree of atrioventricular block (except for pacemaker implantation), systolic blood pressure less than 90mmHg (two vasoactive drugs were already infused continuously )

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The favorable functional outcome of stroke-related disability rate | 90 ± 14 days after thrombectomy
  Modified Rankin Scale ≤ 2 points. mRS range from 0 to 6, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Changes of National Institute of Health stroke scale | 24 ± 6 hours after thrombectomy
  NIHSS (admission) - NIHSS (24h)
Changes of National Institute of Health stroke scale | on the 7-day or discharged day whichever comes first, up to 30 days
  NIHSS (admission) - NIHSS (7day)
Changes of ischemic penumbra | on the 7-day or discharged day whichever comes first, up to 30 days
  The difference of infarct volume between preoperative and 7-day or discharged day
Length of ICU stay | From the date of admission until discharged from ICU, up to 30 days
  Length of ICU stay
Length of hospital stay | From the date of admission until discharged from hospital, up to 30 days
  Length of hospital stay
adverse events at 90-day after operation | within 90-day after thrombectomy
  hypotension (systolic blood pressure under 90mmHg), bradycardia (heart rate under 50bpm), hypoxemia (pulse oxygen saturation under 90%), and serious events such as death and life-threatening events
mortality rate at 90-day after operation | within 90-day after thrombectomy
  Death after thrombectomy within 90-day after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing ChaoYang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and Informed Consent Form will be shared with other researchers.
Supporting Information: Study Protocol, ICF
Time Frame: The information will become available after the publishing of this study and will be available for 1-year after publishing.
Access Criteria: Please contact by E-mail at thoth_safin@sina.com

REFERENCES:
- [Derived] Yang LN, Sun Y, Wang YZ, Wang J, Qi YS, Mu SS, Liu YP, Zhang ZQ, Chen ZM, Wang XJ, Xie WX, Wei CW, Wang Y, Wu AS. Effect of Postoperative Prolonged sedation with Dexmedetomidine after successful reperfusion with Endovascular Thrombectomy on long-term prognosis in patients with acute ischemic stroke (PPDET): study protocol for a randomized controlled trial. Trials. 2024 Mar 4;25(1):166. doi: 10.1186/s13063-024-08015-x. PMID 38439027